CLINICAL TRIAL: NCT04845295
Title: The Effects of Resistance Training on Skeletal Muscle Morphological, Mechanical and Contractile Properties
Brief Title: Resistance Training Effects on Muscle Morphological, Mechanical and Contractile Properties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Vladimir Ilic, Associate Professor, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2316/19-2
Record Dates: First submitted 2021-04-10; First posted 2021-04-14 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Hypertrophy; Contraction
MeSH Terms: conditions — Hypertrophy | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast Tempo (Experimental): Performed training intervention with a tempo of 1 second for eccentric and 1 second for concentric phase
  Interventions: Other: resistance training
- Slow Tempo (Experimental): Performed training intervention with a tempo of 4 seconds for eccentric and 1 second for concentric phase
  Interventions: Other: resistance training

INTERVENTIONS:
Other: resistance training — Both experimental groups performed two exercises to target elbow flexor and knee extensor muscles: biceps curl on a Scott bench and parallel barbell squat, respectively. All sessions were performed at the same time (13-15 h), with a minimum 48 h rest between sessions on the same days during the week. For both groups, the intensity of load (1RM%) and number of sets were as follows: in the first three weeks the subjects exercises with ̴ 60% of 1RM in 3 sets, while during the next four weeks the load was set at ̴ 70% of 1RM in 4 sets. All repetitions were performed until muscular failure. The pause between sets was 2 minutes.

SUMMARY:
The aim of the research project is to investigate the influence of resistance-training prescription (repetition duration, time under tension and training volume) and sex have on morpho-functional adaptations of upper and lower-body skeletal muscles. Twenty-four male and female university students were randomly assigned to one of two experimental groups, based on the repetition duration : "fast" group (with 1 second for eccentric and concentric phase) and "slow" group with prolonged duration of eccentric contraction (4 seconds for eccentric and 1 second concentric phase). At baseline and final measurement, cross-section area, one-repetition maximum and tensiomyography parameters (contraction time - Tc and radial displacement - Dm) of elbow flexors (biceps brachii) and knee extensors (4 quadriceps muscles) were evaluated.

DETAILED DESCRIPTION:
Isotonic resistance training has been widely applied in sport and exercise. Design of resistance training programs depends on numerous training variables, such as intensity, volume, time under tension (TUT), repetition duration (tempo), etc. It has been shown that manipulation of repetition duration affects TUT and training volume, which in turn could results in distinct morphological and contractile adaptative response of skeletal muscle. The aim of the research was three-fold: i) to compare two different tempos of resistance exercise, which differ in the duration of eccentric phase on hypertrophy, strength and contractile properties of the elbow flexors and knee extensors muscles, ii) to compare sex-specific adaptations in hypertrophy, strength and contractile properties of the elbow flexors and knee extensors muscles produced by training intervention, iii) to investigate potential cause-and-effect association between changes in size, strength and contractile properties of the tested muscles.

The subjects were assigned to two experimental groups, based on the duration of the eccentric muscle contraction in resistance training. All participants were fully informed about experimental procedures and potential risks and they signed written informed consent prior to participation in the study. The training intervention was performed twice per week for a 7-week period. Before training intervention, a 2-week familiarization period was conducted. Elbow flexor and knee extensors muscle dimensions and strength were assessed 2 days before and after training intervention, while contractile properties were evaluated 5 days before and after experiment. The number of repetitions, training volume (number of repetitions x number of series), and TUT were recorded after first session of training intervention for both groups.

Muscle strength was assessed by one-repetition maximum test (1RM) for two exercises: elbow flexion on Scott's bench and parallel barbell squat. Each participant had 5 attempts to lift the maximum weight with pauses between trials of 3 minutes.

Muscles cross-section area (CSA) were evaluated by ultrasonic device (Siemens Antares, Erlangen, Germany), using the 2D ellipse diagnostic method with variable high frequency transducer (from 7 MHz to 13 MHz), for 5 muscles: elbow flexor (biceps brachii) and 4 knee extensors (rectus femoris , vastus intermedius, vastus medialis, vastus lateralis). The measurements were performed while the subjects seated with their elbows and knees extended and relaxed. The biceps brachii CSA was measured at two-thirds of the distance from the acromion to the antecubital crease. CSA of rectus femoris was measured at the height of proximal section of its distal third, above musculoskeletal joint. CSA of vastus intermedius and vastus medialis were measured at the height of distal part right above the patella. The visible part of vastus lateralis was measured at the distal third directly above the patella, under rectus femoris level.

The contractile properties of biceps brachii, rectus femoris and vastus lateralis muscles were evaluated by tensiomyography according to the manufacturer's instructions (TMG-Science for Body Evaluation, Ljubljana, Slovenia). The values of contraction time (Tc) and radial deformation (Dm) were taken for analysis. The biceps brachii testing was performed while subjects were in a sitting position with the dominant arm bent at 90°. During the assessment of the knee extensors subjects were lying on the back, where dominant leg was placed on the support, forming a knee angle of 120°. Subjects were asked to perform a voluntary contraction, in order to mark the point of placement of the TMG sensor by the palpation method. Two self-adhesive electrodes (Pals Platinum, model 895220 with multi-stick gel, AxelGaard Manufacturing Co. Ltd) were placed proximal and distal at 3 cm from the marked point, emitting an electrical impulse. A sensor (GK40, Panoptik d.o.o., Ljubljana, Slovenia) was placed between the electrodes to detect muscle changes initiated by electrical stimulation. The initial impulse was 25 milliamperes (mA) and it increased proportionally by 10 mA, until the maximum (muscle no longer responds to electrical stimulus).

Both experimental groups performed two exercises to target elbow flexor and knee extensor muscles: biceps curl on a Scott bench and parallel barbell squat, respectively. All sessions were performed at the same time (13-15 h), with a minimum 48 h rest between sessions on the same days during the week. For both groups, the intensity of load (1RM%) and number of sets were as follows: in the first three weeks the subjects exercises with ̴ 60% of 1RM in 3 sets, while during the next four weeks the load was set at ̴ 70% of 1RM in 4 sets. The difference in training protocols was in the duration of the eccentric phase, where one group performed training with a tempo of 1 seconds for eccentric and concentric phase, while for other group tempo was 4 seconds for eccentric and 1 seconds for concentric phase. All repetitions were performed until muscular failure. The pause between sets was 2 minutes.

Prior to analysis data were checked for normality and that the relevant assumptions for each test were met. Differences in the training volume and the TUT between the groups were determined by an independent t-test. One-way ANCOVA (using baseline values as covariates) was used to examine differences in changes of CSA, 1RM and TMG parameters between the groups. If ANCOVA showed statistical significance, the bonferroni post-hoc test was used for further estimation of differences between groups. Additionally, using sex as between-group factor and baseline values as covariates, ANCOVA was used to determine possible differences between males and females in changes of morphological, mechanical and contractile variables. Relative changes for each variable was derived from Pre to Post change in percentage, and for each participant. Pearson's correlation coefficient was used to examine the association between relative pre-to-post changes of CSA, 1RM and TMG for tested muscles. Data were reported as mean ± standard deviation. The level of significance was set at p < 0.05. The program used for statistical analysis was Statistical Package for Social Sciences (IBM SPSS Statistics), version 20.0.

ELIGIBILITY:
Inclusion Criteria:

* without resistance training participation in past 8 months

Exclusion Criteria:

* history of upper or lower body musculoskeletal injuries

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
muscle hypertrophy | 7 weeks
  cross-section area assessment
muscle strength changes | 7 weeks
  one-repetition maximum assessment
contractile properties changes | 7 weeks
  TMG assessment

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Ilic, Principal Investigator — Faculty of Sport and Physical Education, University of Belgrade
Locations (1):
- Faculty of Sport and Physical Education, Belgrade, Serbia

REFERENCES:
- [Background] Hackett DA, Davies TB, Orr R, Kuang K, Halaki M. Effect of movement velocity during resistance training on muscle-specific hypertrophy: A systematic review. Eur J Sport Sci. 2018 May;18(4):473-482. doi: 10.1080/17461391.2018.1434563. Epub 2018 Feb 12. PMID 29431597
- [Background] Schoenfeld BJ. The mechanisms of muscle hypertrophy and their application to resistance training. J Strength Cond Res. 2010 Oct;24(10):2857-72. doi: 10.1519/JSC.0b013e3181e840f3. PMID 20847704
- [Background] Davies TB, Kuang K, Orr R, Halaki M, Hackett D. Effect of Movement Velocity During Resistance Training on Dynamic Muscular Strength: A Systematic Review and Meta-Analysis. Sports Med. 2017 Aug;47(8):1603-1617. doi: 10.1007/s40279-017-0676-4. PMID 28105573
- [Background] Pisot R, Narici MV, Simunic B, De Boer M, Seynnes O, Jurdana M, Biolo G, Mekjavic IB. Whole muscle contractile parameters and thickness loss during 35-day bed rest. Eur J Appl Physiol. 2008 Sep;104(2):409-14. doi: 10.1007/s00421-008-0698-6. Epub 2008 Feb 23. PMID 18297302
- [Background] Pryor RR, Sforzo GA, King DL. Optimizing power output by varying repetition tempo. J Strength Cond Res. 2011 Nov;25(11):3029-34. doi: 10.1519/JSC.0b013e31820f50cb. PMID 21881531
- [Derived] Kojic F, Mandic D, Ilic V. Resistance training induces similar adaptations of upper and lower-body muscles between sexes. Sci Rep. 2021 Dec 6;11(1):23449. doi: 10.1038/s41598-021-02867-y. PMID 34873221